CLINICAL TRIAL: NCT04207359
Title: The THRIVE Study: An Open-Label Randomized Trial of Exercise ± Creatine Supplementation to Augment the Adaptations of Exercise Training in Breast Cancer Survivors
Brief Title: Effects of Creatine Supplementation in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: ThriveWell Cancer Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTMS# 19-0028; HSC20190610H (Other: UT Health Science Center San Antonio IRB)
Record Dates: First submitted 2019-12-16; First posted 2019-12-20 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Chemotherapy Effect; Muscle Weakness; Muscle Loss; Exercise
Keywords: Special Populations; Exercise Oncology; Creatine Supplementation; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Breast Neoplasms; Muscle Weakness; Muscular Atrophy; Motor Activity | interventions — Creatine

STUDY DESIGN:
Intervention Model Description: This study plans to enroll 30 breast cancer patients who have completed chemotherapy within 6 months prior to consenting for this study. Patients eligible to participate in this study will be allocated to either the creatine group or the control group (1:1) based on a pre-determined randomization list. Each arm will have 15 participants. One arm will receive creatine and the other will serve as the control group with no creatine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Creatine Supplement Group (Experimental): Participants will engage in three center-based exercise sessions each week for 12 weeks; each session lasting roughly 1-hour. Participants will be given a fitbit (electronic watch that measures steps or heart rate) as well to track heart rate and monitor activity throughout the study.
  Interventions: Dietary Supplement: Creatine
- Exercise Only Control Group (No Intervention): Participants will not participate in the creatine intervention (creatine supplementation). Participants will engage in three center-based exercise sessions each week for 12 weeks; each session lasting roughly 1-hour. Exercise sessions will be held by trained study staff held at the Medical Arts and Research Center Physical Therapy clinic (address listed above).

INTERVENTIONS:
Dietary Supplement: Creatine — Those randomized to receive creatine (experimental group) will be initially dosed at 20 g/day for 7 days to boost availability of creatine systemically. Thereafter, the dose will be reduced to 5 g/day for maintenance through the duration of the 12-week protocol.
  Arms: Creatine Supplement Group

SUMMARY:
The purpose of this study is to test the hypothesis that creatine will accelerate adaptations associated with exercise in breast cancer survivors recently completing chemotherapy.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effects of creatine supplementation in modulating strength and physical function in breast cancer survivors that have recently completed chemotherapy. The primary hypothesis for this objective is that creatine will lead to significantly greater gains in strength and physical function in breast cancer survivors compared to exercise alone. The secondary objective is to determine if supplemental creatine can increase intramuscular storage of creatine and alter energy storage. The hypothesis for this objective is that creatine supplementation will significantly increase intramuscular concentrations of creatine (Cr), phosphocreatine (PCr) and adenosine triphosphate (ATP) in the vastus lateralis (VL) compared to controls. The secondary hypothesis for this objective is that the creatine group will have significantly greater muscle cross-sectional area and significantly lower intramuscular fat compared to controls. The final objective for this study is to test the hypothesis that creatine supplementation will improve body composition in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years of age
* Recent (within 6 months) completion of chemotherapy
* Willing to attend 3 virtual exercise sessions per week
* Able to take oral medications
* Participant is willing and able to provide consent to participating in the study
* Serum creatinine ≤ 1.5 x ULN or Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration equation.

Exclusion Criteria:

* Physical indications where performing exercise may be limited and/or contraindicated
* Poorly-controlled hypertension (blood pressure > 160/95mmHg)
* Current tobacco use (within 6 months)
* Anabolic steroids use
* Pitting edema
* Currently undergoing chemotherapy
* History of moderate-severe heart disease (New York Heart Classification greater than grade II) or pulmonary disease (dyspnea on exertion upon climbing one flight of stairs or less; abnormal breath sounds on auscultation).
* Pregnant or plan to get pregnant during the study
* Recent (within one month) or anticipated treatment with corticosteroids (except for short term use during the time of chemotherapy), androgens, progestational agents, or other appetite stimulants
* Serum creatinine > 1.5 x ULN or Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration equation.
* Currently taking creatine supplements

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Change in strength in breast cancer survivors | From baseline to 12 weeks
  Participants will be evaluated for knee extensor strength via isometric maximum voluntary contraction at approximately 60° knee flexion.
Change in functional capacity in breast cancer survivors | From baseline to 12 weeks
  Functional exercise capacity will be assessed via the 6 minute walk test (6MWT).

SECONDARY OUTCOMES:
Change in intramuscular creatine and altering energy storage. | From baseline to 12 weeks
  Muscle Creatine, Phosphocreatine, and Adenosine-triphosphate content will be assessed in vivo by 31P-MRS using a whole body 3.0T MRI scanner.
Change in muscle cross sectional area | From baseline to 12 weeks
  Magnetic resonance imaging will be used to capture the mid-thigh cross section.

CONTACTS AND LOCATIONS:
Overall Officials: Darpan I Patel, PhD, Principal Investigator — UT Health San Antonio
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel DI, Gonzalez A, Moon C, Serra M, Bridges PB, Hughes D, Clarke G, Kilpela L, Jiwani R, Musi N. Exercise and Creatine Supplementation to Augment the Adaptation of Exercise Training Among Breast Cancer Survivors Completing Chemotherapy: Protocol for an Open-label Randomized Controlled Trial (the THRIVE Study). JMIR Res Protoc. 2022 Apr 1;11(4):e26827. doi: 10.2196/26827. PMID 35363152